CLINICAL TRIAL: NCT06946524
Title: A Phase 1 Pharmacokinetic Study in Healthy Subjects to Evaluate the Bioavailability of Risankizumab Following Subcutaneous Administration With Prefilled Pen Relative to Prefilled Syringe
Brief Title: A Study to Assess the Bioavailability of Risankizumab Following Subcutaneous Administration With Prefilled Pen Relative to a Prefilled Syringe in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: M25-681
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Risankizumab
MeSH Terms: interventions — risankizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Risankizumab Arm A (Experimental): Participants will receive a single Subcutaneous (SC) injection of risankizumab Dose A administered via Prefilled Syringe (PFS) at Day 1
  Interventions: Drug: Risankizumab
- Risankizumab Arm B (Experimental): Participants will receive a single Subcutaneous (SC) injection of risankizumab Dose B administered via Prefilled Pen (PFP) at Day 1
  Interventions: Drug: Risankizumab

INTERVENTIONS:
Drug: Risankizumab — Subcutaneous Injection
  Other Names: SKYRIZI

SUMMARY:
This study will assess the pharmacokinetics, relative bioavailability, immunogenicity, safety, and tolerability of risankizumab following subcutaneous (SC) administration with a prefilled pen or a prefilled syringe in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) ≥ 18.0 to ≤ 32.0 kg/m^2 after rounding to the tenths decimal at the time of screening and upon initial confinement. BMI is calculated as weight in kg divided by the square of height measured in meters.
* Body weight greater than 40 kg and less than 100 kg at screening and upon initial confinement.
* A condition of general good health, based upon the results of a medical history, physical examination, vital signs, laboratory profile, and a 12-lead ECG

Exclusion Criteria:

* Previous exposure to any anti-interleukin-12/23 or anti interleukin-23 treatment for at least one year prior to Screening.
* Intention to perform strenuous exercise to which the participant is unaccustomed within one week prior to administration of first dose of study drug and during the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2025-05-08 (Actual); Primary Completion 2025-11-25 (Actual); Study Completion 2025-11-25 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Risankizumab | Up to approximately 141 days
  Maximum observed plasma concentration (Cmax) of Risankizumab
Time to Cmax (Tmax) of Risankizumab | Up to approximately 141 days
  Tmax of Risankizumab
Apparent Terminal Phase Elimination Rate Constant (β) of Risankizumab | Up to approximately 141 days
  Apparent terminal phase elimination rate constant (β) of Risankizumab
Terminal Phase Elimination Half-life (t1/2) of Risankizumab | Up to approximately 141 days
  Terminal phase elimination half-life (t1/2) of Risankizumab
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to the Last Measurable Concentration (AUCt) of Risankizumab | Up to approximately 141 days
  AUCt of Risankizumab
Area Under the Plasma Concentration-Time Curve (AUC) From Time 0 to Infinity (AUCinf) of Risankizumab | Up to approximately 141 days
  AUCinf of Risankizumab
Number of Participants Experiencing Adverse Events | Up to approximately 141 days
  An adverse event is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - Altasciences Clinical Los Angeles /ID# 276446, Cypress, California
  - Acpru /Id# 275116, Grayslake, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M25-681